CLINICAL TRIAL: NCT01050439
Title: Unrelated Donor Stem Cell Transplant for Patients With Malignant and Non-Malignant Disorders
Brief Title: Unrelated Donor Transplant for Malignant and Non-Malignant Disorders
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PI left the institution
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAB3095; CHNY-02-516 (Other: CU)
Record Dates: First submitted 2008-06-03; First posted 2010-01-15 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Leukemia; Lymphoma; Bone Marrow Failure Syndromes; Immunodeficiencies; Histiocytosis
Keywords: Allogeneic Stem Cell Transplant; Unrelated donor; Cord blood donor
MeSH Terms: conditions — Leukemia; Lymphoma; Bone Marrow Failure Disorders; Immunologic Deficiency Syndromes; Histiocytosis | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- UDAlloSCT + Therapy (Experimental): This is a non-randomized study to test the safety and response of unrelated matched donor allogeneic stem cell transplantation (UDAlloSCT) with either myleoablative (full intensity) or reduced intensity conditioning therapy in patients with selected malignant and non-malignant disorders. UDAlloSCT has been performed in both adults and children as an alternative transplant for patients who lack and HLA-matched family donor in both malignant and non-malignant disease with varying degrees of response.
  Interventions: Procedure: UDAlloSCT; Other: Therapy

INTERVENTIONS:
Procedure: UDAlloSCT — unrelated matched donor allogeneic stem cell transplantation (UDAlloSCT)
Other: Therapy — Full Intensity Therapy (myeloablative) (TBI + Thiotepa + Cyc) OR Reduced Intensity Therapy (Fludarabine, Busulfan, and Alemutuzumab (FBA))

SUMMARY:
Unrelated matched donor (cord blood, bone marrow or peripheral blood) allogeneic stem cell transplantation (UDAlloSCT) with either myeloablative or reduced intensity conditioning will be well tolerated and result in a high degree of engraftment in patients with selected malignant and non malignant disorders.

DETAILED DESCRIPTION:
This is a non-randomized study to determine the tolerability and degree of engraftment of unrelated matched donor allogeneic stem cell transplantation with either myeloablative or reduced intensity conditioning in patients with selected malignant and non malignant disorders. Patients will receive one of either full intensity or reduced intensity regimen based on the patient's disease status, organ function and performance and determined by the PI.

ELIGIBILITY:
Inclusion Criteria:

* Adequate renal function defined as: serum creatinine 2.0 x normal, or creatinine clearance or radioisotope GFR > 40 ml/min/m2 or > 40 ml/min/1.73 m2 or an equivalent GFR as determined by the institutional normal range.
* Adequate liver function defined as: total bilirubin < 2.5 x normal; or SGOT (AST) or SGPT (ALT) < 5.0 x normal.
* Adequate cardiac function defined as: shortening fraction of > 25% by echocardiogram, or ejection fraction of > 40% by radionuclide angiogram or echocardiogram.
* Adequate pulmonary function defined as: DLCO > 35% by pulmonary function test. For children who are uncooperative, no evidence of dyspnea at rest, no exercise intolerance, and a pulse oximetry > 94% in room air.
* Diseases:

  * CML (CP, AP or BC)
  * AML/MDS/JCML
  * ALL
  * Lymphoma (Hodgkin's and non-Hodgkin's)
  * Non-malignant disorders
* Bone Marrow Failure Syndromes: Patients with the following diagnoses are eligible:

  * Severe Aplastic Anemia:
  * Fanconi Anemia
  * Severe Congenital Neutropenia (Kostmann's Syndrome)
  * Amegakaryocytic Thrombocytopenia
  * Diamond-Blackfan Anemia
  * Infantile Osteopetrosis
  * Schwachman-Diamond Syndrome
  * Dyskeratosis Congenita
  * Other bone marrow failure syndromes at discretion of Principal Investigator
* Immunodeficiencies:

  * SCIDS, all subtypes
  * Combined Immunodeficiency Syndrome
  * Wiskott-Aldrich syndrome
  * Chronic Granulomatous Disease
  * Chediak-Higashi Syndrome
  * Leukocyte Adhesion Deficiency
  * Other immunodeficiencies at discretion of Principal Investigator
* Inborn Errors of Metabolism (IEOM):

  * Transplant is recommended for the following disorders: Hurler syndrome (L-iduronidase deficiency, MPS-I), Maroteaux-Lamy syndrome (galactosamine-4-sulfatase deficiency, MP VI), Sly syndrome (glucuronidase deficiency, MPS-VII), Globoid cell Leukodystrophy (galactocerebrosidasedeficiency), Metachromatic leukodystrophy (arylsulfatase A deficiency), Childhood-onset X-linked adrenoleukodystrophy (X-ALD), Fucosidosis (fucosidase deficiency), Mannosidosis, Aspartylglucosaminuria, Niemann-Pick Disease Type B (acid sphingomyelinase deficiency), Gaucher disease (glucocerebrosidase deficiency) Type I (non neuropathic), Other diagnoses may be considered at the discretion of the Principal Investigator
  * For X-ALD patients greater than 5 years of age, IQ > 80 is required. For other patients greater than 5 years of age, IQ > 70 is required.
  * For patients less than 5 years of age, the developmental quotient or clinical neurodevelopmental examination should demonstrate potential for stabilization at a level of functioning where continuous life support (e.g. mechanical ventilation) would not be predicted to be required in the year following transplantation.
* Histiocytosis:

  * Hemophagocytic Lymphohistiocytosis (HLH)
  * Familial Erythrophagocytic Lymphohistiocytosis
  * Langerhans Cell Histiocytosis
  * Malignant Histiocytosis
* Other Malignant and non-malignant diseases: Other malignant and non-malignant diseases not listed above may be eligible if deemed appropriate by the Principal Investigator.

Exclusion Criteria:

* Women who are pregnant and/or breast feeding are ineligible

Max Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2002-11; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Incidence of toxicity related to myeloablative therapy | Up to 10 years from start of study
  To determine the safety and toxicity of myeloablative therapy (TBI + Melphalan) and unrelated donor alloSCT in selected patients with malignant and non-malignant disorders.

SECONDARY OUTCOMES:
Incidence of toxicity related to reduced intensity therapy | Up to 10 years from start of study
  To determine the safety and toxicity of reduced intensity therapy (Fludarabine, Busulfan, and Alemtuzumab (FBA) and unrelated donor alloSCT in selected patients with malignant and non malignant disorders
Percentage of donor chimerism | Up to 10 years from start of study
  To quantitate the percentage of donor chimerism following both myeloablative and reduced intensity conditioning and unrelated donor alloSCT in selected patients with malignant and non-malignant disorders.
Prevalence of progression free survival | Up to 10 years from start of study
  To estimate the progression free survival (PFS), if applicable, event free survival (EFS) and overall survival (OS) following unrelated donor alloSCT in selected patients with malignant and non malignant disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell S Cairo, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States